CLINICAL TRIAL: NCT06896344
Title: Microenvironment Cross-talk: Role of Extracellular Vesicles Derived From Mesenchymal Stromal Cells of Patients With Primary Myelofibrosis in Modifying Functional Activities of CD34+ Hematopoietic Progenitor Cells
Brief Title: Role of Mesenchymal Stromal Cell Derived Extracellular Vesicles of Primary Myelofibrosis Patients on CD34+ Cells
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Margherita Massa, Principal investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: Microenvironment cross-talk; 08052022 (Other: Ministry of Health)
Record Dates: First submitted 2025-03-06; First posted 2025-03-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Primary Myelofibrosis
Keywords: Primary Myelofibrosis; CD34; extracellular vesicles
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will retain extracellular vescicle (EV) samples. Evs may contain smal amount of DNA, RNA, proteins, lipids, all derived from the parental cell
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with PMF out of therapy undergoing bone marrow biopsy for clinical reasons: Healthy subjects who donate bone marrow hematopoietic progenitor cells
  Interventions: Other: In vitro culture

INTERVENTIONS:
Other: In vitro culture — In vitro culture of bone marrow MNCs to obtain mesenchymal stromal cells

SUMMARY:
The aim of this study is to demonstrate that, in patients with myelofibrosis (PMF), a chronic neoplastic disease of the bone marrow, some of the cells that form the bone marrow microenvironment (mesenchymal stromal cells, MSCs) can send wrong messages to the CD34+ hematopoietic progenitor cells (HPCs). CD34+ HPCs in normal conditions reside in the bone marrow until complete maturation; in PMF they leave the bone marrow when they are still progenitor cells and frequently they express the V617F mutation on the JAK2 molecule. In previously published papers, the investigators demonstrated that the MSCs in the bone marrow of patients with PMF are different from those in healthy donors. In this study the investigators want to verify how this difference affects the maturation of CD34+ HPCs of healthy donors and of SET2 cells, a commercially available cell line characterized by the V617F mutation of the JAK2 molecule. In particular, the investigators will verify the effect of MSCs on signals that induce the activation of CD34+ cells, their survival or death, the production of harmful oxidative reagents and their clonal capacity. To obtain these data, the investigators will isolate MSCs from bone marrow blood samples of patients with PMF undergoing bone marrow biopsy for clinical reasons and from healthy subjects, donors of HPCs for transplant. Following a long culture MSCs will be stimulated to release small vescicles containing part of their nuclear and cytoplasmatic molecules. These vescicles will be cultured with CD34+ cells or SET2 cells and their effects will be evaluated. It has been shown that these small vescicles act exactly like MSCs, but they are easier to be used, and could become a very useful acellular drug in the near future.

DETAILED DESCRIPTION:
Primary myelofibrosis (PMF) is a chronic myeloproliferative neoplasm characterized by the clonal proliferation of CD34+ progenitor cells. A constitutive activation of the JAK-STAT pathway, due to an acquired gain of function mutation either in JAK2, MPL or CALR genes, plays a relevant pathogenetic role. Moreover, a state of chronic inflammation affects the disease course. Currently, the therapy with the JAK inhibitor Ruxolitinib ameliorates the symptoms of the disease, with no effects on the pathological cell clone; hematopoietic progenitor cell (HPC) transplantation is the only curative option. The investigators previously published that mesenchymal stromal cells (MSCs) from patients with PMF display functional and genetic abnormalities (low proliferative potential, precocious senescence, reduced differentiation potential). Regarding Ruxolitinib, direct effects on MSCs have been described, such as the inhibition of the JAK-STAT signaling, the growth of both healthy donor (HD)- and PMF-MSCs, and the decrease of fibrosis related gene expression. Ruxolitinib has also been reported to reduce MSC secretion of inflammatory cytokines MCP-1 and IL-6, suggesting a role of this drug in modifying the bone marrow (BM) microenvironment. In PMF, as in other hematological malignancies, MSCs participate in the communication between microenvironment and CD34+ cells. Recent studies demonstrated in other pathologies that MSC-derived extracellular vesicles (EVs) and parental MSCs have similar effects. In fact EVs, containing mRNA, microRNA, lipids, and proteins can be incorporated into recipient cells and modify their functions. In normal hematopoiesis, MSC-EV incorporation in CD34+ cells has been shown to induce an activation of the JAK-STAT pathway through increased levels of phospho-STAT5; in addition, a significant decrease in apoptosis and a higher colony-forming unit granulocyte/macrophage clonogenic potential have been reported.

The objectives of this study are:

* to isolate MSCs from BM of PMF patients and HDs. MSCs will be incubated with/out Ruxolitinib. EVs will be obtained following MSC starvation and ultracentrifugations, and stored at -80°C
* to assess EV effects on HD-CD34+ or JAK2V617F+ SET2 cells by evaluation of apoptotic and activation pathways, ROS production and clonogenic capacity. To this regard, confirmatory experiments will be performed with JAK2-mutated CD34+ cells from patients receiving or not Ruxolitinib.
* to perform gene expression profile on CD34+ and SET2 cells after incubation with EVs.
* to investigate EV biocargoes both qRT-PCR and proteomics will be performed on MSC-derived EVs, before and after incubation with Ruxolitinib.

The expected impact will include the identification of modifications in functional activities of CD34+ or SET2 cells following incubation with PMF-MSC-EVs with respect to HD-MSC-EVs, reflecting the effect of an altered microenvironment on HPCs. The investigators also expect the recognition of important targets of severity/progression of the disease by assessing the gene expression profile in CD34+ or SET2 cells that incorporate EVs from different sources.

In addition, the identification of the Ruxolitinib effects on PMF BM microenvironment may be clarified.

This study may allow to act on new targets of disease progression or to support the future use of HD-EVs as an acellular therapy that favours the survival of healthy CD34+ cells or acts against their clonal counterpart.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PMF
* JAK2 V617F+ (either homozygous or heterozygous)
* Out of therapy
* At least 18 years old

Exclusion Criteria:

* PMF combined to other pathologies
* Previous splenectomy
* Previous bone marrow transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PMF (WHO 2016) afferent at the Center for the Study of Myelofibrosis, a national center that receives patients from all the country. Patients will be out of therapy, undergoing bone marrow biopsy for clinical reasons.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Effect of bone marrow microenvironment, resembled by EVs, on hematopoietic progenitor cells | Up to 24 weeks
  The measure of the functional activities of HD-CD34+ cells induced by the bone marrow microenvironment (i.e. MSC derived EVs) of patients with PMF or heathy donors. P-STAT5 molecule as activation index, Bax/Bcl2 ratio as apoptosis indicator, ROS and membrane antigens will be assessed by a unique unit of measure, the mean fluorescence intensity. The change of the different parameters from baseline to the end of the co-culture will be reported.

SECONDARY OUTCOMES:
Components of EV biocargoes | Through study completion, an average of 1 year
  Molecular analysis of EV biocargoes derived from either PMF or healthy MSCs

CONTACTS AND LOCATIONS:
Overall Officials: Margherita Massa, PhD, Principal Investigator — IRCCS Policlinico San Matteo Foundation
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zacharaki D, Ghazanfari R, Li H, Lim HC, Scheding S. Effects of JAK1/2 inhibition on bone marrow stromal cells of myeloproliferative neoplasm (MPN) patients and healthy individuals. Eur J Haematol. 2018 Jul;101(1):57-67. doi: 10.1111/ejh.13079. Epub 2018 Apr 30. PMID 29645296
- [Background] Preciado S, Muntion S, Corchete LA, Ramos TL, de la Torre AG, Osugui L, Rico A, Espinosa-Lara N, Gastaca I, Diez-Campelo M, Del Canizo C, Sanchez-Guijo F. The Incorporation of Extracellular Vesicles from Mesenchymal Stromal Cells Into CD34+ Cells Increases Their Clonogenic Capacity and Bone Marrow Lodging Ability. Stem Cells. 2019 Oct;37(10):1357-1368. doi: 10.1002/stem.3032. Epub 2019 Jun 11. PMID 31184411